CLINICAL TRIAL: NCT02103127
Title: Evaluation of the Picosure 755nm Alexandrite Laser With Lens Array for the Treatment of Acne Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN13-PCAP-AS-SK02
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Acne Scars
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm Alexandrite laser with lens array (Experimental)
  Interventions: Device: 755nm Alexandrite laser with lens array

INTERVENTIONS:
Device: 755nm Alexandrite laser with lens array

SUMMARY:
The purpose of this study is to assess treatment of facial acne scars using the 755nm Alexandrite Laser with lens arrays.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female between 18 and 65 years old
2. Has unwanted acne scars, excluding ice pick scars (Deep atrophic scars that resemble poked holes), and wishes to undergo laser treatments.
3. Is willing to consent to participate in the study.
4. Is willing to comply with all requirements of the study including biopsies, being photographed, following post treatment care and attending all treatment and follow up visits.

Exclusion Criteria:

1. The subject is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
2. The subject is hypersensitive to light exposure OR takes photo sensitized medication.
3. The subject has active or localized systemic infections.
4. The subject has a coagulation disorder or is currently using anti-coagulation medication (including but not limited to heavy aspirin therapy {greater than 81 mg per day}).
5. The subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within 3 months prior to entering this study.
7. The subject has used Accutane within 6 months prior to enrollment.
8. The subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.
9. The subject has had prior treatment with parenteral gold therapy (gold sodium thiomalate).
10. The subject has a history of keloids.
11. The subject has evidence of compromised wound healing.
12. The subject has a history of squamous cell carcinoma or melanoma.
13. The subject has a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
14. The subject has an allergy to lidocaine and epinephrine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Laser & Skin Surgery Center of Northern California, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 755nm Alexandrite Laser With Lens Array: 755nm Alexandrite laser with lens array
Period: Overall Study
Arm/Group | 755nm Alexandrite Laser With Lens Array
Started | 20
Completed | 17
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | 755nm Alexandrite Laser With Lens Array
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 16
  Race/Ethnicity: Asian | 0
  Race/Ethnicity: African American | 0
  Race/Ethnicity: Hispanic | 3
  Race/Ethnicity: Other | 1
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Score I | 0
    Fitzpatrick Skin Score II | 13
    Fitzpatrick Skin Score III | 3
    Fitzpatrick Skin Score IV | 4
    Fitzpatrick Skin Score V | 0
    Fitzpatrick Skin Score VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Severity Change in Acne Scarring
Description: The scale is a Physician Global Scarring Grading Scale, which counts and types scars by tallying up of the number and severity according to an organized grading system, where 0 is the lowest point value and represents no scarring. The theoretical highest score possible is an 84. The change in the score from the baseline to the follow up was collected. A negative change indicates a decrease in points (which indicates improvement).
Time Frame: Baseline and 1 month post treatment
Population: 1 subject was pregnant, 1 subject was lost to follow up, and 1 subject withdrew consent. 3 subjects missed their visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser With Lens Array
Number analyzed (Participants) | 14
score on a scale | -2 (2.71)

2. Secondary Outcome: Investigator Satisfaction Questionnaire
Description: Investigator will complete satisfaction questionnaire at follow up visits from 0 to 3, where 0 is extremely dissatisfied and 3 is extremely satisfied.
Time Frame: 3 months post treatment
Population: 1 subject was pregnant, 1 subject was lost to follow up, and 1 subject withdrew consent.
Measure: Number; unit: participants
Arm/Group | 755nm Alexandrite Laser With Lens Array
Number analyzed (Participants) | 17
participants
  Extremely Satisfied | 0
  Satisfied | 10
  Dissatisfied | 7
  Extremely Dissatisfied | 0

3. Secondary Outcome: Subject Satisfaction Questionnaire
Description: Subject will complete satisfaction questionnaire at follow up visits from 0 to 3, where 0 is extremely dissatisfied and 3 is extremely satisfied.
Time Frame: 3 months post treatment
Population: 1 subject was pregnant, 1 subject was lost to follow up, and 1 subject withdrew consent.
Measure: Number; unit: participants
Arm/Group | 755nm Alexandrite Laser With Lens Array
Number analyzed (Participants) | 17
participants
  Extremely Satisfied | 3
  Satisfied | 11
  Dissatisfied | 3
  Extremely Dissatisfied | 0

4. Primary Outcome: Severity Change in Acne Scarring
Description: as for outcome 1
Time Frame: Baseline and 3 months post treatment
Population: 1 subject was pregnant, 1 subject was lost to follow up, and 1 subject withdrew consent.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 755nm Alexandrite Laser With Lens Array
Number analyzed (Participants) | 17
score on a scale | -1 (3.15)

ADVERSE EVENTS:
Time Frame: Adverse Events occurring will be captured and followed throughout each subject's participation in the study, approximately 10 months.
Arm/Group | 755nm Alexandrite Laser With Lens Array
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 17/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 755nm Alexandrite Laser With Lens Array (N=20)
Redness (Skin and subcutaneous tissue disorders) | 17
Edema (Skin and subcutaneous tissue disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.